CLINICAL TRIAL: NCT03320850
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Single-treatment, 2-stage, Dose-finding Study Evaluating the Efficacy and Safety of BOTOX® Intravesical Instillation in Participants With Overactive Bladder and Urinary Incontinence
Brief Title: BOTOX® Intravesical Instillation in Participants With Overactive Bladder and Urinary Incontinence
Acronym: APOLLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839-201-021
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Urinary Incontinence; Overactive Bladder With Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 100U cohort - BOTOX® plus Hydrogel admixture (Experimental): 100U BOTOX® (onabotulinumtoxinA) and Hydrogel admixture administered as a single intravesical instillation on Day 1
  Interventions: Drug: OnabotulinumtoxinA and Hydrogel admixture
- 100U cohort - Placebo plus Hydrogel admixture (Placebo Comparator): Placebo and Hydrogel admixture administered as a single intravesical instillation on Day 1
  Interventions: Drug: Placebo and Hydrogel admixture
- 300U cohort - BOTOX® plus Hydrogel admixture (Experimental): 300U BOTOX® (onabotulinumtoxinA) and Hydrogel admixture administered as a single intravesical instillation on Day 1
  Interventions: Drug: OnabotulinumtoxinA and Hydrogel admixture
- 300U cohort - Placebo plus Hydrogel admixture (Placebo Comparator): Placebo and Hydrogel admixture administered as a single intravesical instillation on Day 1
  Interventions: Drug: Placebo and Hydrogel admixture
- 400U cohort - BOTOX® plus Hydrogel admixture (Experimental): 400U BOTOX® (onabotulinumtoxinA) and Hydrogel admixture administered as a single intravesical instillation on Day 1
  Interventions: Drug: OnabotulinumtoxinA and Hydrogel admixture
- 400U cohort - Placebo plus Hydrogel admixture (Placebo Comparator): Placebo and Hydrogel admixture administered as a single intravesical instillation on Day 1
  Interventions: Drug: Placebo and Hydrogel admixture
- 500U cohort - BOTOX® plus Hydrogel admixture (Experimental): 500U BOTOX® (onabotulinumtoxinA) and Hydrogel admixture administered as a single intravesical instillation on Day 1
  Interventions: Drug: OnabotulinumtoxinA and Hydrogel admixture
- 500U cohort - Placebo plus Hydrogel admixture (Placebo Comparator): Placebo and Hydrogel admixture administered as a single intravesical instillation on Day 1
  Interventions: Drug: Placebo and Hydrogel admixture

INTERVENTIONS:
Drug: OnabotulinumtoxinA and Hydrogel admixture — BOTOX® (onabotulinumtoxinA) and Hydrogel admixture administered as a single intravesical instillation
  Other Names: BOTOX®; Botulinum Toxin Type A
  Arms: 100U cohort - BOTOX® plus Hydrogel admixture; 300U cohort - BOTOX® plus Hydrogel admixture; 400U cohort - BOTOX® plus Hydrogel admixture; 500U cohort - BOTOX® plus Hydrogel admixture
Drug: Placebo and Hydrogel admixture — Placebo and Hydrogel admixture administered as a single intravesical instillation
  Arms: 100U cohort - Placebo plus Hydrogel admixture; 300U cohort - Placebo plus Hydrogel admixture; 400U cohort - Placebo plus Hydrogel admixture; 500U cohort - Placebo plus Hydrogel admixture

SUMMARY:
This study will evaluate the efficacy and safety of BOTOX® intravesical instillation in participants with overactive bladder and urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of OAB (frequency/urgency) with urinary incontinence for at least 6 months
* Inadequate response or limiting side effects with pharmacotherapy for the treatment of OAB

Exclusion Criteria:

* Overactive Bladder caused by neurological condition
* Patient has predominance of stress incontinence
* History or evidence of pelvic or urological abnormality
* Prior use of BOTOX for any urological condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Till Geib, Study Director — Allergan
Locations (63):
- United States (61):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Coastal Clinical Research, Inc., an AMR company, Mobile, Alabama
  - Urological Assoc. of South AZ, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - San Bernardino Urological Associates Medical Group, San Bernardino, California
  - Wr-McCr, Llc, San Diego, California
  - San Diego Clinical Trials, San Diego, California
  - Sutter Institute for Medical Health, Vacaville, California
  - West Coast Urology, Whittier, California
  - The Urology Center of Colorado, Denver, Colorado
  - Urology Associates, P.C, Englewood, Colorado
  - Adult and Pediatric Urology, Bridgeport, Connecticut
  - Women's Health Specialty Care, Farmington, Connecticut
  - CT Clinical Research Center/Urologist Specialist, Middlebury, Connecticut
  - Innovative Medical Research of South FL, Inc., Aventura, Florida
  - South Florida Medical Research, Aventura, Florida
  - Manatee Medical Research Institute, Bradenton, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Urological Research Network, Miramar, Florida
  - Florida Urology Partners, North Redington Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Institute, Meridian, Idaho
  - Comprehensive Urological Care, Lake Barrington, Illinois
  - Urogynecology Associates, PC, Carmel, Indiana
  - First Urology,PSC, Jeffersonville, Indiana
  - The Iowa Clinic, West Des Moines, Iowa
  - DelRicht Research, LLC, New Orleans, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Associates, Hanover, Maryland
  - Chesapeake Urology, Owings Mills, Maryland
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Women's Health Care Specialists, Kalamazoo, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - Adult Pediatric Urology & Urogynecology, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Premier Urology Group, Edison, New Jersey
  - Delaware Valley Urology, Mount Laurel, New Jersey
  - Western New York Urology Associates, Cheektowaga, New York
  - AccuMed Research Associates, Garden City, New York
  - Urological Surgeons of Long Island, Garden City, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Urology Institute of Long Island, Plainview, New York
  - Associated Medical Professionals- Urology, Syracuse, New York
  - American Health Research, Charlotte, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Clinical Research Solutions, LLC, Middleburg Heights, Ohio
  - The Center for Men's & Women's Urology, Gresham, Oregon
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Urology Clinics of North Texas, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Washington Urology and Urogynecology Associates, Kirkland, Washington
  - Multicare Allenmore Hospital, Tacoma, Washington
  - Aurora Research Institute, West Allis, Wisconsin
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
* Phase II or III trials completed after 2008
  * Listed on clinicaltrials.gov or EudraCT
  * Have received regulatory approval in the United States and/or European Union (depending on registration plans) in a given indication
  * Primary manuscript(s) from the trial have been published
  Access to data is contingent upon the following:
  * Researcher signs a data use agreement from Allergan
  * Data is to be used for non-commercial purposes

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. — http://AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: Placebo + Hydrogel Admixture; Stage 2: Placebo + Hydrogel Admixture: BOTOX® matching-placebo and hydrogel admixture administered as a single intravesical instillation on Day 1.
- Stage 1: BOTOX® 100U + Hydrogel Admixture: BOTOX® 100 units (U) (onabotulinumtoxinA; botulinum toxin Type A) and hydrogel admixture administered as a single intravesical instillation on Day 1.
- Stage 1: BOTOX® 300U + Hydrogel Admixture; Stage 2: BOTOX® 300U + Hydrogel Admixture: BOTOX® 300U (onabotulinumtoxinA) and hydrogel admixture administered as a single intravesical instillation on Day 1.
- Stage 1: BOTOX® 400U + Hydrogel Admixture; Stage 2: BOTOX® 400U + Hydrogel Admixture: BOTOX® 400U (onabotulinumtoxinA) and hydrogel admixture administered as a single intravesical instillation on Day 1.
- Stage 1: BOTOX® 500U + Hydrogel Admixture; Stage 2: BOTOX® 500U + Hydrogel Admixture: BOTOX® 500U (onabotulinumtoxinA) and hydrogel admixture administered as a single intravesical instillation on Day 1.
- Stage 2: BOTOX® 100U + Hydrogel Admixture: BOTOX® 100U (onabotulinumtoxinA) and hydrogel admixture administered as a single intravesical instillation on Day 1.
Period: Overall Study
Arm/Group | Stage 1: Placebo + Hydrogel Admixture | Stage 1: BOTOX® 100U + Hydrogel Admixture | Stage 1: BOTOX® 300U + Hydrogel Admixture | Stage 1: BOTOX® 400U + Hydrogel Admixture | Stage 1: BOTOX® 500U + Hydrogel Admixture | Stage 2: Placebo + Hydrogel Admixture | Stage 2: BOTOX® 100U + Hydrogel Admixture | Stage 2: BOTOX® 300U + Hydrogel Admixture | Stage 2: BOTOX® 400U + Hydrogel Admixture | Stage 2: BOTOX® 500U + Hydrogel Admixture
Started | 18 | 12 | 18 | 22 | 19 | 58 | 57 | 60 | 60 | 59
Safety Population (Safety Population included all participants enrolled in this study who received the study treatment in Stage 1 and Stage 2.) | 18 | 12 | 18 | 22 | 19 | 57 | 57 | 60 | 60 | 58
Completed | 18 | 12 | 18 | 21 | 17 | 49 | 50 | 53 | 50 | 50
Not Completed | 0 | 0 | 0 | 1 | 2 | 9 | 7 | 7 | 10 | 9
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 5 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3
Not completed — Failure to Meet Randomization Criteria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Stage 1: Safety Analysis Set included all participants who were randomized and treated; Stage 2: Intent-to-treat (ITT) Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: Placebo + Hydrogel Admixture | Stage 1: BOTOX® 100U + Hydrogel Admixture | Stage 1: BOTOX® 300U + Hydrogel Admixture | Stage 1: BOTOX® 400U + Hydrogel Admixture | Stage 1: BOTOX® 500U + Hydrogel Admixture | Stage 2: Placebo + Hydrogel Admixture | Stage 2: BOTOX® 100U + Hydrogel Admixture | Stage 2: BOTOX® 300U + Hydrogel Admixture | Stage 2: BOTOX® 400U + Hydrogel Admixture | Stage 2: BOTOX® 500U + Hydrogel Admixture | Total
Number analyzed (Participants) | 18 | 12 | 18 | 22 | 19 | 58 | 57 | 60 | 60 | 59 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Stage 1: Safety Analysis Set included all participants who were randomized and treated.
  years
    number analyzed (Participants) | 18 | 12 | 18 | 22 | 19 | 0 | 0 | 0 | 0 | 0 | 89
    (all) | 55.7 (13.8) | 54.7 (13.0) | 56.2 (12.1) | 62.4 (8.6) | 55.3 (13.2) |  |  |  |  |  | 57.2 (12.2)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Stage 2: Intent-to-treat (ITT) Analysis Set included all randomized participants.
  years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 58 | 57 | 60 | 60 | 59 | 294
    (all) |  |  |  |  |  | 57.9 (11.17) | 60.4 (9.93) | 59.1 (11.33) | 59.8 (9.10) | 60.7 (9.38) | 59.6 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 15 | 18 | 17 | 53 | 53 | 54 | 54 | 54 | 347
  Male | 1 | 0 | 3 | 4 | 2 | 5 | 4 | 6 | 6 | 5 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 1 | 0 | 5 | 9 | 5 | 11 | 7 | 45
  Not Hispanic or Latino | 16 | 10 | 15 | 21 | 19 | 53 | 48 | 55 | 49 | 52 | 338
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 1 | 7 | 12 | 13 | 10 | 9 | 16 | 80
  White | 13 | 8 | 14 | 20 | 11 | 44 | 44 | 48 | 49 | 43 | 294
  More than one race | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Stage 1: Average Number of Urinary Incontinence Episodes (UIE) [Mean (Standard Deviation); unit: episodes per day] — The participant recorded urinary incontinence (lack of voluntary control over urination) in a 3-day bladder diary. The average number of urinary incontinence episodes per day is the average of the 3-day diary entries. Population: Safety Analysis Set included all participants who were randomized and treated in Stage 1.
  episodes per day
    number analyzed (Participants) | 18 | 12 | 18 | 22 | 19 | 0 | 0 | 0 | 0 | 0 | 89
    (all) | 7.1 (3.4) | 4.7 (2.5) | 5.8 (2.7) | 4.4 (2.7) | 5.3 (3.0) |  |  |  |  |  | 5.5 (3.0)
Stage 2: Average Number of Urinary Incontinence Episodes [Mean (Standard Deviation); unit: episodes per day] — The participant recorded urinary incontinence (lack of voluntary control over urination) in a 3-day bladder diary. The average number of urinary incontinence episodes per day is the average of the 3-day diary entries. Population: ITT Analysis Set included all randomized participants in Stage 2. Overall number analyzed is the number of participants with data available for analyses at the Baseline.
  episodes per day
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 57 | 57 | 60 | 60 | 59 | 293
    (all) |  |  |  |  |  | 6.06 (3.162) | 5.60 (4.267) | 4.46 (2.738) | 4.56 (3.073) | 5.92 (3.302) | 5.30 (3.386)
Stage 1: Average Number of Micturition Episodes per Day [Mean (Standard Deviation); unit: episodes per day] — The participant recorded the number of micturition (urination in toilet or catherization) episodes per day in a 3-day bladder diary. The average number of micturition episodes per day is the average of the 3-day diary entries. Population: Safety Analysis Set included all participants who were randomized and treated in Stage 1.
  episodes per day
    number analyzed (Participants) | 18 | 12 | 18 | 22 | 19 | 0 | 0 | 0 | 0 | 0 | 89
    (all) | 10.6 (2.4) | 10.9 (3.5) | 10.0 (1.6) | 11.3 (2.4) | 11.8 (2.9) |  |  |  |  |  | 10.9 (2.6)
Stage 2: Average Number of Micturition Episodes per Day [Mean (Standard Deviation); unit: episodes per day] — The participant recorded the number of micturition (urination in toilet or catherization) episodes per day in a 3-day bladder diary. The average number of micturition episodes per day is the average of the 3-day diary entries. Population: ITT Analysis Set included all randomized participants in Stage 2. Overall number analyzed is the number of participants with data available for analyses at the Baseline.
  episodes per day
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 57 | 57 | 60 | 60 | 59 | 293
    (all) |  |  |  |  |  | 11.12 (3.049) | 10.97 (2.938) | 10.91 (2.678) | 9.88 (2.030) | 10.70 (2.822) | 10.71 (2.738)
Stage 1: Average Volume Voided per Micturition [Mean (Standard Deviation); unit: milliliter (mL)] — Volume voided per micturition was recorded over one 24-hour period during the 3-day bladder diary. Population: Safety Analysis Set included all participants who were randomized and treated in Stage 1.
  milliliter (mL)
    number analyzed (Participants) | 18 | 12 | 18 | 22 | 19 | 0 | 0 | 0 | 0 | 0 | 89
    (all) | 189.2 (64.1) | 189.8 (94.0) | 182.5 (79.3) | 150.0 (54.7) | 199.4 (70.0) |  |  |  |  |  | 180.4 (71.9)
Stage 2: Average Volume Voided per Micturition [Mean (Standard Deviation); unit: mL] — Volume voided per micturition was recorded over one 24-hour period during the 3-day bladder diary. Population: ITT Analysis Set included all randomized participants in Stage 2. Overall number analyzed is the number of participants with data available for analyses at the Baseline.
  mL
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 57 | 57 | 60 | 60 | 59 | 293
    (all) |  |  |  |  |  | 179.10 (59.421) | 173.28 (66.615) | 167.10 (67.940) | 194.50 (67.414) | 199.58 (74.154) | 182.79 (68.025)

OUTCOME MEASURES:

1. Primary Outcome: Stage 2: Change From Baseline in the Average Number of Urinary Incontinence Episodes (UIEs) Per Day
Description: The participant recorded urinary incontinence (lack of voluntary control over urination) in a 3-day bladder diary. The average number of UIEs per day is the average of the 3-day diary entries. A negative change from Baseline indicates improvement. Baseline is defined as the last non-missing assessment before the first dose of study treatment. An analysis of covariance (ANCOVA) model was used for analyses.
Time Frame: Baseline (3 consecutive days during Day -14 to Day -1) to 3 consecutive days in the Week prior to Week 12
Population: Participants from the Intent-to-treat (ITT) Analysis Set, all randomized participants in Stage 2, with data available for analysis at Baseline and Week 12. As per protocol, this endpoint is only applicable to the Stage 2 arms.
Measure: Least Squares Mean (Standard Error); unit: episodes per day
Arm/Group | Stage 2: Placebo + Hydrogel Admixture | Stage 2: BOTOX® 100U + Hydrogel Admixture | Stage 2: BOTOX® 300U + Hydrogel Admixture | Stage 2: BOTOX® 400U + Hydrogel Admixture | Stage 2: BOTOX® 500U + Hydrogel Admixture
Number analyzed (Participants) | 57 | 57 | 60 | 60 | 58
episodes per day | -2.72 (0.534) | -1.62 (0.539) | -0.89 (0.521) | -1.52 (0.520) | -1.85 (0.530)
Statistical Analysis 1: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 100U + Hydrogel Admixture; The null hypothesis is that there is no difference between each (BOTOX® and Hydrogel admixture group) and (placebo and Hydrogel admixture) in the mean change from Baseline in daily average number of UIEs at Week 12; Test type: Superiority; p = 0.0845, ANCOVA; Least Squares Mean Difference = 1.10, 95% CI 2-sided [-0.15 to 2.35], Standard Error of Mean 0.635 — Least square estimates and contrast t-test were used to compare specified treatment groups and were based on ANCOVA model with Baseline value as covariate and treatment group, sex (male, female) as factors
Statistical Analysis 2: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 300U + Hydrogel Admixture; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0041, ANCOVA; Least Squares Mean Difference = 1.83, 95% CI 2-sided [0.59 to 3.08], Standard Error of Mean 0.633 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 400U + Hydrogel Admixture; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0600, ANCOVA; Least Squares Mean Difference = 1.19, 95% CI 2-sided [-0.05 to 2.44], Standard Error of Mean 0.632 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 500U + Hydrogel Admixture; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1702, ANCOVA; Least Squares Mean Difference = 0.87, 95% CI 2-sided [-0.37 to 2.11], Standard Error of Mean 0.631 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAEs) in the Treatment Period
Description: An adverse event (AE) is any untoward medical occurrence in a participants or clinical study investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. A TEAE is an AE that occurs or worsens after receiving study drug.
Time Frame: Up to End of Study (Stage 1: Up to 114 days and Stage 2: Up to 35.1 weeks)
Population: Safety Analysis Set included all randomized and treated participants in Stages 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Placebo + Hydrogel Admixture | Stage 1: BOTOX® 100U + Hydrogel Admixture | Stage 1: BOTOX® 300U + Hydrogel Admixture | Stage 1: BOTOX® 400U + Hydrogel Admixture | Stage 1: BOTOX® 500U + Hydrogel Admixture | Stage 2: Placebo + Hydrogel Admixture | Stage 2: BOTOX® 100U + Hydrogel Admixture | Stage 2: BOTOX® 300U + Hydrogel Admixture | Stage 2: BOTOX® 400U + Hydrogel Admixture | Stage 2: BOTOX® 500U + Hydrogel Admixture
Number analyzed (Participants) | 18 | 12 | 18 | 22 | 19 | 57 | 57 | 60 | 60 | 58
Participants | 6 | 4 | 4 | 10 | 6 | 25 | 30 | 30 | 38 | 25

3. Secondary Outcome: Stage 2: Change From Baseline in the Average Number of Micturition Episodes Per Day
Description: The participant recorded the number of micturition (urination in toilet or catherization) episodes per day in a 3-day bladder diary. The average number of micturition episodes per day is the average of the 3-day diary entries. A negative change from Baseline indicates improvement. Baseline is defined as the last non-missing assessment before the first dose of study treatment. ANCOVA model was used for analyses.
Time Frame: Baseline (3 consecutive days during Days -14 to Day -1) to 3 consecutive days in the Week prior to Week 12
Population: Participants from the ITT Analysis Set, all randomized participants in Stage 2, with data available for analysis at Baseline and Week 12. As per protocol, this endpoint is only applicable to the Stage 2 arms.
Measure: Least Squares Mean (Standard Error); unit: episodes per day
Arm/Group | Stage 2: Placebo + Hydrogel Admixture | Stage 2: BOTOX® 100U + Hydrogel Admixture | Stage 2: BOTOX® 300U + Hydrogel Admixture | Stage 2: BOTOX® 400U + Hydrogel Admixture | Stage 2: BOTOX® 500U + Hydrogel Admixture
Number analyzed (Participants) | 46 | 49 | 52 | 55 | 52
episodes per day | -1.64 (0.519) | -0.91 (0.514) | -0.86 (0.486) | -1.00 (0.480) | -1.11 (0.492)
Statistical Analysis 1: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 100U + Hydrogel Admixture; Test type: Superiority; p = 0.2361, ANCOVA; Least Square Mean = 0.73, 95% CI 2-sided [-0.48 to 1.95], Standard Error of Mean 0.617 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 300U + Hydrogel Admixture; Test type: Superiority; p = 0.1985, ANCOVA; Least Square Mean = 0.78, 95% CI 2-sided [-0.41 to 1.98], Standard Error of Mean 0.608 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 400U + Hydrogel Admixture; Test type: Superiority; p = 0.2923, ANCOVA; Least Square Mean = 0.64, 95% CI 2-sided [-0.56 to 1.84], Standard Error of Mean 0.607 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 500U + Hydrogel Admixture; Test type: Superiority; p = 0.3769, ANCOVA; Least Square Mean = 0.54, 95% CI 2-sided [-0.66 to 1.74], Standard Error of Mean 0.609 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Stage 2: Change From Baseline in the Average Volume Voided Per Micturition
Description: Volume voided per micturition was recorded over one 24-hour period during the 3-day bladder diary. The volume voided during each 24-hour period was divided by the number of micturitions during the period. The average volume voided per micturition is the average of the 3-day diary entries. A negative change from Baseline indicates improvement. Baseline is defined as the last non-missing assessment before the first dose of study treatment. ANCOVA model was used for analyses.
Time Frame: Baseline (3 consecutive days during Days -14 to Day -1) to 3 consecutive days in the Week prior to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Stage 2: Placebo + Hydrogel Admixture | Stage 2: BOTOX® 100U + Hydrogel Admixture | Stage 2: BOTOX® 300U + Hydrogel Admixture | Stage 2: BOTOX® 400U + Hydrogel Admixture | Stage 2: BOTOX® 500U + Hydrogel Admixture
Number analyzed (Participants) | 46 | 49 | 52 | 55 | 51
mL | 12.61 (11.251) | 5.56 (11.214) | 4.61 (10.576) | 11.28 (10.349) | 21.94 (10.779)
Statistical Analysis 1: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 100U + Hydrogel Admixture; Test type: Superiority; p = 0.5911, ANCOVA; Least Square Mean = -7.05, 95% CI 2-sided [-32.87 to 18.77], Standard Error of Mean 13.107 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 300U + Hydrogel Admixture; Test type: Superiority; p = 0.5375, ANCOVA; Least Square Mean = -8.00, 95% CI 2-sided [-33.52 to 17.52], Standard Error of Mean 12.956 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 400U + Hydrogel Admixture; Test type: Superiority; p = 0.9173, ANCOVA; Least Square Mean = -1.33, 95% CI 2-sided [-26.47 to 23.81], Standard Error of Mean 12.764 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Stage 2: Placebo + Hydrogel Admixture vs Stage 2: BOTOX® 500U + Hydrogel Admixture; Test type: Superiority; p = 0.4730, ANCOVA; Least Square Mean = 9.33, 95% CI 2-sided [-16.24 to 34.90], Standard Error of Mean 12.981 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to End of Study (Stage 1: Up to 114 days and Stage 2: Up to 35.1 weeks)
Description: All-Cause Mortality: ITT Analysis Set included all randomized participants. Serious Adverse Events and Other Adverse Events: Safety Analysis Set included all randomized and treated participants in Stages 1 and 2.
Arm/Group | Stage 1: Placebo + Hydrogel Admixture | Stage 1: BOTOX® 100U + Hydrogel Admixture | Stage 1: BOTOX® 300U + Hydrogel Admixture | Stage 1: BOTOX® 400U + Hydrogel Admixture | Stage 1: BOTOX® 500U + Hydrogel Admixture | Stage 2: Placebo + Hydrogel Admixture | Stage 2: BOTOX® 100U + Hydrogel Admixture | Stage 2: BOTOX® 300U + Hydrogel Admixture | Stage 2: BOTOX® 400U + Hydrogel Admixture | Stage 2: BOTOX® 500U + Hydrogel Admixture
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12 | 0/18 | 0/22 | 0/19 | 0/58 | 0/57 | 0/60 | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12 | 0/18 | 0/22 | 0/19 | 1/57 | 3/57 | 1/60 | 2/60 | 0/58
Other Adverse Events (participants affected / at risk) | 6/18 | 4/12 | 4/18 | 4/22 | 6/19 | 10/57 | 17/57 | 17/60 | 16/60 | 19/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Placebo + Hydrogel Admixture (N=18) | Stage 1: BOTOX® 100U + Hydrogel Admixture (N=12) | Stage 1: BOTOX® 300U + Hydrogel Admixture (N=18) | Stage 1: BOTOX® 400U + Hydrogel Admixture (N=22) | Stage 1: BOTOX® 500U + Hydrogel Admixture (N=19) | Stage 2: Placebo + Hydrogel Admixture (N=57) | Stage 2: BOTOX® 100U + Hydrogel Admixture (N=57) | Stage 2: BOTOX® 300U + Hydrogel Admixture (N=60) | Stage 2: BOTOX® 400U + Hydrogel Admixture (N=60) | Stage 2: BOTOX® 500U + Hydrogel Admixture (N=58)
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Stage 1: Placebo + Hydrogel Admixture (N=18) | Stage 1: BOTOX® 100U + Hydrogel Admixture (N=12) | Stage 1: BOTOX® 300U + Hydrogel Admixture (N=18) | Stage 1: BOTOX® 400U + Hydrogel Admixture (N=22) | Stage 1: BOTOX® 500U + Hydrogel Admixture (N=19) | Stage 2: Placebo + Hydrogel Admixture (N=57) | Stage 2: BOTOX® 100U + Hydrogel Admixture (N=57) | Stage 2: BOTOX® 300U + Hydrogel Admixture (N=60) | Stage 2: BOTOX® 400U + Hydrogel Admixture (N=60) | Stage 2: BOTOX® 500U + Hydrogel Admixture (N=58)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Instillation site discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 3 | 3 | 1 | 2 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 5 | 8 | 8 | 4 | 9
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 2 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 0/17 | 0 | 0/15 | 1/18 | 0/17 | 0/53 | 0/53 | 0/54 | 0/54 | 0/54 — Number of participants at risk are Female participants as this adverse event is specific to Females.
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 4
Acetonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 5
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 2
Urethral pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03320850/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03320850/SAP_001.pdf